CLINICAL TRIAL: NCT06739785
Title: Turkish Translation And Cross-Cultural Adaptation of The Sport Concussion Assessment Tool 6th Edition (SCAT6)
Brief Title: Turkish Translation of SportsConcussion Assesment Tool 6
Acronym: SCAT 6-tr
Status: Active, not recruiting | Type: Observational
Sponsor: Ordu University (Other)
Collaborators: Ankara Medipol University (Other)
Responsible Party: Principal Investigator, FUAT YUKSEL, Principal Investigator, Ordu University
Other Study IDs: E-1467249-000-1071258
Record Dates: First submitted 2024-12-13; First posted 2024-12-18 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2024-12

CONDITIONS: Sports Injury; Concussion, Mild; Concussion, Brain; Concussion, Severe; Concussion, Intermediate
MeSH Terms: conditions — Athletic Injuries; Brain Concussion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: SCAT6-tr — Step 1: Initial Translation At this stage, two independent bilingual translators whose native language is Turkish will translate the content into Turkish. Step 2: Integration of Translations
  A single translation will be created by comparing the two Turkish versions of SCAT 6.
  Step 3: Back-translation The Turkish version will be translated into English by 2 bilingual colleagues who are blind to the original version. The Turkish version will be translated into English by 2 bilingual colleagues who are blind to the original version. These two English versions will be compared, differences will be resolved by consensus and a new combined version will be created. If consensus cannot be reached, a third person will be asked for help. Step 4: Expert Evaluation

SUMMARY:
Concussions, a significant type of sports injury caused by head, face, or neck trauma, are common in contact sports and require serious attention due to potential fatal consequences of mismanagement. The Sport Concussion Assessment Tool (SCAT), developed by the Concussion in Sport Group (CISG) and updated in 2023, provides a standardized approach to assess head injuries and manage athletes' return-to-sport process. While SCAT has been adapted into various languages, no Turkish version exists. This study aims to translate and culturally adapt SCAT 6 into Turkish, contributing to the accurate evaluation and management of concussion injuries among Turkish-speaking athletes.

DETAILED DESCRIPTION:
Concussions constitute an important part of sports injuries. Concussion is a head trauma caused by blows to the head, face and neck. Head injuries are common in contact sports. They are usually minor injuries. However, injuries should be taken seriously. Because mismanagement can be fatal in cases of misdiagnosis. Therefore, it is among medical emergencies .

A sports concussions group has been established for the correct management of concussions seen in sports. In 2022, the group met in Amsterdam, renewed the existing consensus and published it in the British Journal of Sports Medicine in 2023 . The Sport Concussion Assessment Tool (SCAT), developed by the sports concussion group (CISG), is a valid and reliable approach to assessing sports-related head injuries ('Sport Concussion Assessment Tool 6 (SCAT6),' 2023). The main purpose of SCAT is to assess head injuries with a standardised method and to manage the return to sport process of athletes. SCAT is an assessment tool that evaluates adult athletes over the age of 13 in terms of physical, mental and cognitive aspects and includes different sections.

In the literature, there are adaptations of previous and current versions of SCAT in different languages (Korean, Chinese, Persian, Arabic). However, no Turkish translation and adaptation study of any version has been conducted before. Turkishisation of this assessment tool is an important step in terms of accurately evaluating concussion injuries in Turkish-speaking athletes and managing the return to sport process correctly. The aim of this study is to translate the SCAT 6 into Turkish and to provide intercultural adaptation of the SCAT 6 to the literature.

ELIGIBILITY:
Inclusion Criteria:

To be 13 years old

* Talking in Turkish
* Being a Professional Athlete

Exclusion Criteria:

* Athletes who experience any injury during the test, retest process will be excluded from the study.

Min Age: 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Athletes
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-09-15 (Actual); Primary Completion 2025-11-15 (Estimated); Study Completion 2025-12-15 (Estimated)

PRIMARY OUTCOMES:
Lawshe Analysis | Before the create last verison of SCAT6-tr .It is planned to take 1 month.
  The appropriateness of the assessment tool will be determined by analysing the expert opinion forms reported by the experts.

SECONDARY OUTCOMES:
Inter-rater reliability | After the last version created. It is planned to take 2 months
  Scat 6-Tr will be applied randomly to 30 athletes by 2 different assessors. Scat 6-Tr will be applied randomly to 30 athletes by 2 different assessors. Inter-rater correlation will be analysed by Intra-class Correlation Coefficient (ICC).
Test-retest reliability. | After the last version created. It is planned to take 2 months
  SCAT6-tr will be administered to 30 athletes 2 times by the same assessor at 1 week intervals. The correlation between measurements will be evaluated with Intra-class Correlation Coefficient (ICC).

CONTACTS AND LOCATIONS:
Locations (1):
- Ordu University, Ordu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No